CLINICAL TRIAL: NCT04416880
Title: Effectiveness of Press Tack Needle Acupuncture in Treating Lactation Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Diana Oei, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medical Acupuncture 2019
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Lactation; Insufficient, Partial; Hypogalactia, Without Mention of Attachment Difficulty
Keywords: acupuncture; exclusive breastfeeding; breastmilk; press tack needle; lactation insufficiency
MeSH Terms: conditions — Breast Feeding; Lactation Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Press Tack Needle Acupuncture (Experimental): Patients in this group were given seirin pyonex press tack needle treatment in the acupuncture points CV17 Danzhong and SI1 Shaoze bilateral for 7 days.
  Interventions: Device: Press Tack Needle Acupuncture
- Sham Control Press Tack Needle Acupuncture (Sham Comparator): Patients in this group were given sham treatment in the acupuncture points CV17 Danzhong and SI1 Shaoze bilateral for 7 days.
  Interventions: Device: Press Tack Needle Acupuncture

INTERVENTIONS:
Device: Press Tack Needle Acupuncture — Seirin Pyonex Press Tack Needle 0.20 x 0.60 mm for SI1 Shaoze acupuncture point Seirin Pyonex Press Tack Needle 0.20 x 0.90 mm for CV17 Danzhong acupuncture point

SUMMARY:
This study was meant to see the effectiveness of press tack needle acupuncture in improving lactation insufficiency. The acupuncture points used in this study were CV17 Danzhong and SI1 Shaoze. Press Tack Needles were placed in these acupuncture points for 7 days in hope that it will give continuous acupuncture stimulation that might help in improving lactation insufficiency with minimal side effect, less time consuming, and more efficient for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Breastfeeding mother who suffers from lactation insufficiency
* Breastfeeding mother from 2 weeks to 5 months post-partum
* Breastfeeding mother with healthy baby

Exclusion Criteria:

* Subject consumes drugs that are known to decrease breastmilk production
* Subject with infection or inflammation in the intended acupuncture points
* Subject with bleeding disorder
* Subject consumes anticoagulant
* Subject with known diabetic history
* Subject with body temperature > 38 degree celcius

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Breastfeeding mothers
Enrollment: 36 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Breastmilk Volume | Day 7 of acupuncture or sham treatment
  Pre- and Post Treatment Breastmilk Volume were measured using electric breast pump
Breastmilk Volume | Day 10 of acupuncture or sham treatment (Day 3 after press tack needles were removed)
  Pre- and Post Treatment Breastmilk Volume were measured using electric breast pump

CONTACTS AND LOCATIONS:
Overall Officials: Diana Oei, MD, Principal Investigator — Faculty of Medicine University of Indonesia
Locations (3):
- Indonesia (3):
  - Puskesmas Kecamatan Menteng, Jakarta Pusat, DKI Jakarta
  - Poliklinik Akupunktur Medik RSCM, Jakarta Pusat, DKI Jakarta
  - Puskesmas Kelurahan Pegangsaan, Jakarta Pusat, DKI Jakarta

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR